CLINICAL TRIAL: NCT05952011
Title: Effect of Stellate Ganglion Block on Internal Mammary Artery Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Diaaeldin Badr Aboelnile, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD124/2023
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The first group (A) Stellate Ganglion Block Group (Experimental): Participants in this group will receive a left stellate ganglion block (LSGB) preoperatively. The IMA pulsatility index and diameter will be measured before and after the stellate ganglion block and during both the preoperative and the intraoperative periods. Transit-time flowmetry (TTFM) will be used intraoperatively to assess IMA flow.
  Interventions: Procedure: Left stellate ganglion block; Drug: Topical Nitroglycerine
- The second Group (B) Control Group (No left stellate ganglion block LSGB) (Active Comparator): Participants in this group will not receive a stellate ganglion block. The IMA pulsatility index and diameter will be measured before and after the stellate ganglion block and during both the preoperative and the intraoperative periods. Transit-time flowmetry (TTFM) will be used intraoperatively to assess IMA flow. Topical nitroglycerin will also be applied intraoperatively, similar to the SGB group.
  Interventions: Drug: Topical Nitroglycerine

INTERVENTIONS:
Procedure: Left stellate ganglion block — patients will be positioned with head in midline position and mild extension of the neck. Cricoid cartilage will be identified by midline palpation of the neck and a 12 mega hertz ultrasound probe will be used. The airway will be identified by the shadow of the cricoid cartilage at the level of C6 vertebrae. The probe will be moved laterally to identify internal jugular vein, carotid artery and thyroid. Depth of ultrasound field will be adjusted to include the transverse process of the C6 vertebra. Following complete aseptic precautions, an echogenic insulated needle 5 cm long will be inserted under ultrasound guidance and directed toward the transverse process of the C6 vertebra. After the needle tip will make contact with the transverse process, it will be withdrawn 2 mm and 8 ml of 0.25% bupivacaine will be injected.
  Arms: The first group (A) Stellate Ganglion Block Group
Drug: Topical Nitroglycerine — Application of topical Nitroglycerin solution to the LIMA pedicle graft during dissection of the vessel in both study arms.

SUMMARY:
This study aims to assess the effect of a stellate ganglion block on the flow and diameter of the internal mammary artery using the pulsatility index and transient time flowmetry(TTFM) in patients undergoing coronary artery bypass grafting.

DETAILED DESCRIPTION:
The internal mammary artery (IMA) is the preferred graft for myocardial revascularization because of its superiority over venous grafts owing to long term patency, lower mortality rates and improved post-operative outcomes.

However, conduit spasm is a recognized complication of coronary artery bypass surgery mainly affecting the arterial conduits, a major concern that can lead to acute myocardial ischemia and may contribute to reduce graft patency.

Topical application or systemic administration of many pharmacological agents has been shown to reverse or prevent graft spasm, but side effects are reported with the use of these agents.

Various vasodilators that have been tried included various organic nitrates, calcium channel blockers, sodium nitroprusside (SNP) and papaverine.

Over the last few years, there were some studies, which investigated the effect of regional anesthesia techniques such as thoracic epidural anesthesia (TEA) and stellate ganglion block (SGB) for sympatholysis and studied its effects on internal mammary artery diameter .

The stellate ganglion block with local anesthetics have been widely used to provide pain relief to treat vascular spastic disorders of upper limbs, chronic pain conditions and treatment of refractory angina.

The stellate ganglion block has also been used for increasing radial artery (RA) blood flow and preventing RA spasm by sympathetic blockade in coronary artery bypass surgery.

In our study, two groups will be compared regarding IMA blood flow and diameter. The IMA pulsatility index and diameter will be measured before and after the stellate ganglion block during both the preoperative and intraoperative periods in both groups. Transit-time flowmetry (TTFM) will be used intraoperatively to assess IMA flow. Additionally, topical nitroglycerin will be applied intraoperatively in both groups, regardless of whether they received the stellate ganglion block.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years.
* Patients who will be slated to undergo elective coronary artery bypass graft surgery under Cardiopulmonary bypass in the Department of Cardiothoracic Surgery.

Exclusion Criteria:

* Patient not willing to participate in the study.
* Age more than 65 years.
* Ejection fraction < 45%.
* History of strokes / Transient ischaemic attacks and vertebro basilar insufficiency
* History of Glaucoma.
* History of allergy to local anaesthetic drugs.
* Emergency coronary artery bypass graft or reoperations.
* Pre-existing contralateral phrenic nerve palsy.
* Patients with existing coagulopathy.
* Allergy to nitroglycerin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Effect of left stellate ganglion block on the left internal mammary artery blood flow after 10 minutes | 10 minutes after the left Stellate Ganglion Block
  LIMA blood flow will be measured using the pulsatility index

SECONDARY OUTCOMES:
Change in Left Internal Mammary Artery (LIMA) diameter after left Stellate Ganglion Block | 10 minutes after block
  LIMA diameter measurement using ultrasound
Effect of left stellate ganglion block on the left internal mammary artery blood flow after cardiopulmonary bypass | After cardiopulmonary bypass
  Measurement of LIMA blood flow using transit time flow measurement.
Effect of left stellate ganglion block on mean blood pressure (MBP) | During surgery: baseline, after induction of anesthesia, at time after skin incision, after sternotomy, before and after cardiopulmonary bypass (CPB), after protamine and at the end of operation
  Effect of the block on hemodynamics
Effect of left stellate ganglion block on heart rate (HR)) | During surgery: baseline, after induction of anesthesia, at time after skin incision, after sternotomy, before and after cardiopulmonary bypass (CPB), after protamine and at the end of operation
  Effect of the block on hemodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Diaaeldin DA Aboelnile, MD, Lecturer, Principal Investigator — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No